CLINICAL TRIAL: NCT01223885
Title: Camel's Milk as a Safe Alternative in Cow's Milk Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM-MK-2
Record Dates: First submitted 2010-10-10; First posted 2010-10-19 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2012-08

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Camel's milk, Cow's milk allergy (Experimental)
  Interventions: Dietary Supplement: Camel's milk

INTERVENTIONS:
Dietary Supplement: Camel's milk — Patients with proved cow's milk allergy who have negative prick skin tests to came's milk will be administered gradually increased doses of pasteurized camel's milk at 30 minute intervals

SUMMARY:
By performing a challenge with camel's milk in patients who are allergic to cow's milk, the investigators will examine if camel's milk is a safe alternative for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Proved cow"s milk allergy

Exclusion Criteria:

* Pregnant women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Development of allergic symptoms after graded oral challenge with camel's milk | 3 hours follow-up after completion of the challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Allergy Unit, Meir Medical Center, Kfar Saba, Israel